CLINICAL TRIAL: NCT00366067
Title: Randomised, Placebo Controlled, Double Blind, Parallel Group 3-Months Study of Phenytoin Efficacy in Children for Therapy of Bronchial Asthma
Brief Title: Study of Efficacy of Phenytoin in Therapy of Children With Bronchial Asthma
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Centre of Chinese Medicine, Georgia (Other)
Collaborators: Rea Rehabilitation Centre, Georgia (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LTPZ-P-CH-0806-0107
Record Dates: First submitted 2006-08-17; First posted 2006-08-18 (Estimated); Last update posted 2009-02-19 (Estimated); Status verified 2009-02

CONDITIONS: Bronchial Asthma
Keywords: Bronchial asthma; Phenytoin; Antiepileptic drugs; Efficacy
MeSH Terms: conditions — Asthma | interventions — Phenytoin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Phenytoin

SUMMARY:
The purpose of this study was to determine whether antiepileptic drug phenytoin is effective in the treatment of chronic asthma in children.

DETAILED DESCRIPTION:
Effective therapy of asthma still remains quite serious problem. According GINA definition, asthma is an inflammatory disorder. Consequently, modern pharmacotherapy of asthma provides wide use of anti-inflammatory drugs. But asthma also is a paroxysmal disorder: many specialists and even some guidelines underline paroxysmal clinical picture of asthma. Besides this, according to some authors, neurogenic inflammation may play important role in asthma mechanism. It is known that some other neurogenic inflammatory paroxysmal disorders exist, and they are migraine and trigeminal neuralgia. Antiepileptic drug phenytoin is very effective in therapy of trigeminal neuralgia - more than in 70-80% of cases. Other antiepileptic drugs, salts of valproic acid, are effective in the treatment of migraine. If bronchial asthma also is paroxysmal inflammatory disease, like migraine and trigeminal neuralgia, it is possible that some antiepileptic drugs also are very effective in asthma therapy.

We perform a double-blind, placebo-controlled 3-month trial for evaluation of phenytoin efficacy in therapy of bronchial asthma in children. Phenytoin is a well-known, comparatively safe and effective antiepileptic drug with low cost. According our previous data, phenytoin is effective drug for asthma therapy in adults.

Comparison: children will receive investigational drug in addition to their usual routine antiasthmatic treatment, compared to patients received placebo in addition to their usual routine antiasthmatic treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Patients between 10 and 14, patients parents or supervisors must have given their informed consent before commencing the procedures specified in the protocol, indicating that they understand the objectives of the study and are willing to adhere to the procedures described in the protocol.
2. Patients able to use peak flow meters, to perform spirometry and to swallow capsules.
3. Patient aged between 4 and 14 years, males or females.
4. Out patients.
5. Patients with an established (i.e. at least 6 months) clinical history of asthma.
6. Absence of long-term remissions of asthma (lasting more than 1 month)
7. Poorly controlled asthma, due to various reasons.

Exclusion Criteria:

1. History or presence of cardiovascular, renal, neurologic, psychiatric, liver, immunologic, endocrine, infection or other diseases or dysfunctions if they are clinically significant. A clinically significant disease is defined as one which in the opinion of the investigator may either put the patient at risk because of participation in the study or a disease which may influence the results of the study or the patient's ability to participate in the study.
2. Patients with active tuberculosis with indication for treatment.
3. Patients with clinically significant abnormal baseline haematology, blood chemistry or urinalysis or if the abnormal defines a disease listed as an exclusion criterion.
4. Patients with known allergy, side effects, intolerance/hypersensitivity to investigational drug
5. Patients currently using MAO inhibitors, tricyclic antidepressants, antiepileptic drugs, narcotic agents.
6. Patients between 10 and 14, parents or supervisor of patients unlikely, unable or unwilling to comply with the requirements of the protocol.

Ages: 4 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50
Dates: Start 2006-08; Study Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
At 3 months of treatment: Change from baseline of the FEV1 and PEFR (also %predicted); Number of patients without asthma symptoms

SECONDARY OUTCOMES:
At 3 months of treatment: Difference in PEF pm-am (in %); The daily (daytime and night-time) symptoms scores; % of symptom free days during the treatment period; Use of other antiasthmatic medication

CONTACTS AND LOCATIONS:
Overall Officials: Merab Lomia, MD, PhD, Principal Investigator — "Rea" Rehabilitation Centre; Tamuna Tchelidze, Principal Investigator — CRO Evidence; Nana Zhorzholadze, MD, Principal Investigator — "Rea" Rehabilitation Centre; Manana Pruidze, Study Director — Centre of Chinese Medicine
Locations (1):
- "Rea" Rehabilitation Centre, Tbilisi, Georgia

REFERENCES:
- See also: Bronchial asthma as neurogenic paroxysmal inflammatory disorder — http://www.asthma.ge
- See also: Bronchial asthma as neurogenic paroxysmal inflammatory disease: a randomized trial with carbamazepine — http://www.ncbi.nlm.nih.gov/pubmed/16597501?ordinalpos=2&itool=EntrezSystem2.PEntrez.Pubmed.Pubmed_ResultsPanel.Pubmed_DefaultReportPanel.Pubmed_RVDocSum